CLINICAL TRIAL: NCT01070784
Title: An Open-label Phase III, Multi-centre 52-week , Parallel-group Study Evaluating the Safety and Efficacy of Symbicort Turbuhaler 320/9 Twice Daily Compared With Standard Treatment in Japanese Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Safety and Efficacy Study of Symbicort Turbuhaler Compared With Standard Chronic Obstructive Pulmonary Disease (COPD) Treatment in Japan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D589DC00008
Record Dates: First submitted 2010-02-11; First posted 2010-02-18 (Estimated); Results first posted 2013-12-05 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Symbicort; Safety; Efficacy; COPD; Japanese
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide, Formoterol Fumarate Drug Combination; Budesonide; Formoterol Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Symbicort Turbuhaler (Budesonide/formoterol)
- 2 (Active Comparator)
  Interventions: Drug: Drug: any available COPD treatment; investigator to decide

INTERVENTIONS:
Drug: Symbicort Turbuhaler (Budesonide/formoterol) — 2 x 160/4.5 microgram, inhalation, bid, 52 weeks
  Other Names: Symbicort Turbuhaler
  Arms: 1
Drug: Drug: any available COPD treatment; investigator to decide — According to investigator decision, 52 weeks, Standard COPD treatment according to investigator decision
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Symbicort Turbuhaler compared to standard COPD treatment during one year in Japanese patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* A current clinical diagnosis of COPD according to the guidelines (GOLD, JPS)
* Documented COPD symptoms for more than 2 years
* Pre-bronchodilator FEV1≦50% of predicted normal value, and post-bronchodilator FEV1/FVC<70%

Exclusion Criteria:

* History and/or current clinical diagnosis of asthma and atopic diseases such as allergic rhinitis
* Subjects with significant or unstable ischemic heart disease, arrhythmia, cardiomyopathy, heart failure, uncontrolled hypertension as defined by the investigator, or any other relevant cardiovascular disorder as judged by the investigator
* COPD exacerbation during the run-in period or within 4 weeks prior to registration, requiring hospitalization and/or treatment with systemic steroids.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Andersson, MD, Study Chair — AstraZeneca, R&D, Lund, Sweden
Locations (17):
- Japan (17):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Toyota, Aichi-ken
  - Research Site, Yanagawa, Fukuoka
  - Research Site, Hiroshima, Hiroshima
  - Research Site, Asahikawa, Hokkaido
  - Research Site, Sapporo, Hokkaido
  - Research Site, Itami, Hyōgo
  - Research Site, Hitachi, Ibaraki
  - Research Site, Tsukuba, Ibaraki
  - Research Site, Sakaidechō, Kagawa-ken
  - Research Site, Fujisawa, Kanagawa
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kōshi, Kumamoto
  - Research Site, Kyoto, Kyoto
  - Research Site, Murata, Miyagi
  - Research Site, Chūō, Tokyo
  - Research Site, Setagaya City, Tokyo

REFERENCES:
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=397&filename=CSR-D589DC00008.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first participant entered the study on 28 January 2010, and the last participant completed the study on 24 October 2011. A total of 328 participants were enrolled at 60 centres in Japan, and 260 participants who fulfilled the randomisation criteria were randomised.
Pre-assignment Details: The study starts with an enrolment visit, Visit 1 prior to any other study-related activity. At Visit 2, the lung function will be measured to assess the eligibility of the patients. Subjects who fulfil all eligibility criteria will begin the 2-week run-in period.During the period, the previous treatment will be continued to record the baseline.
Groups:
- Symbicort Turbuhaler: Symbicort Turbuhaler, 160/4.5 microgram(mcg), 2 inhalations twice daily
- COPD Standard Therapy: Standard COPD treatment according to JRS guideline and GOLD guideline
Period: Overall Study
Arm/Group | Symbicort Turbuhaler | COPD Standard Therapy
Started | 130 | 130
Completed | 110 | 112
Not Completed | 20 | 18
Not completed — Withdrawal by Subject | 6 | 9
Not completed — Adverse Event | 14 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort Turbuhaler | COPD Standard Therapy | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Continuous [Mean (Full Range); unit: Years] | 70.1 [40 to 87] | 71.5 [54 to 85] | 70.8 [40 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 125 | 126 | 251

OUTCOME MEASURES:

1. Primary Outcome: Clinical Laboratory Test: Haematology -Erythrocytes
Description: Mean change from Baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: *10000/μl
Groups:
- Arm 1 - Symbicort Turbuhaler: Symbicort Turbuhaler, 160/4.5 microgram(mcg), 2 inhalations twice daily
- Arm 2 - COPD Standard Therapy: Standard COPD treatment according to JRS guideline and GOLD guideline
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 120
*10000/μl | -7.6 (23.9) | -0.1 (22.9)

2. Primary Outcome: Clinical Laboratory Test: Haematology -Haemoglobin
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 120
g/dL | -0.22 (0.74) | -0.05 (0.75)

3. Primary Outcome: Clinical Laboratory Test: Haematology -Leucocytes
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: /microliter(mcl)
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 123 | 120
/microliter(mcl) | 160.8 (1704.0) | -184.8 (1238.2)

4. Primary Outcome: Clinical Laboratory Test: Haematology -Platelet Count
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: *10000/μl
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 120 | 117
*10000/μl | 0.86 (3.03) | 0.12 (4.04)

5. Primary Outcome: Clinical Laboratory Test: Haematology -Eosinophils
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: percentage of Eosinophils
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 123 | 120
percentage of Eosinophils | -0.52 (2.68) | 0.14 (1.91)

6. Primary Outcome: Clinical Laboratory Test: Haematology -Basophils
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: percentage of Basophils
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 123 | 120
percentage of Basophils | -0.06 (0.37) | -0.06 (0.35)

7. Primary Outcome: Clinical Laboratory Test: Haematology -Lymphocytes
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: percentage of Lymphocytes
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 123 | 120
percentage of Lymphocytes | -5.47 (6.56) | -3.24 (7.00)

8. Primary Outcome: Clinical Laboratory Test: Haematology -Monocytes
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: percentage of Monocytes
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 123 | 120
percentage of Monocytes | 0.29 (1.41) | -0.03 (1.35)

9. Primary Outcome: Clinical Laboratory Test: Haematology -Neutrophils
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: percentage of Neutrophils
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 111 | 97
percentage of Neutrophils | 5.78 (7.16) | 2.92 (7.64)

10. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-Alanine Aminotransferase
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
U/L | 0.5 (7.6) | 1.5 (6.6)

11. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-Aspartate Aminotransferase
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
U/L | 0.0 (7.6) | 1.1 (6.5)

12. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-Alkaline Phosphatase (ALP)
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
U/L | 1.3 (38.4) | 8.2 (45.9)

13. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-Creatinine
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
mg/dL | 0.003 (0.106) | -0.017 (0.091)

14. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-Total Bilirubin
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
mg/dL | 0.05 (0.25) | 0.00 (0.18)

15. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-Sodium
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
mEq/L | -0.8 (2.0) | -0.6 (1.7)

16. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-Potassium
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
mEq/L | -0.11 (0.34) | -0.08 (0.37)

17. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S- Calcium
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
mg/dL | 0.02 (0.34) | 0.01 (0.33)

18. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-Albumin
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
g/dL | 0.03 (0.24) | 0.04 (0.26)

19. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-Protein, Total
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
g/dL | 0.01 (0.35) | 0.02 (0.37)

20. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-C-Reactive Protein
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
mg/dL | 0.243 (1.291) | 0.224 (1.423)

21. Primary Outcome: Clinical Laboratory Test: Clinical Chemistry- S-Urea Nitrogen
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 124 | 119
mg/dL | -0.51 (4.09) | -0.64 (3.32)

22. Primary Outcome: Vital Signs- Sitting Systolic Blood Pressure(SBP)
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 126 | 125
mmHg | -0.8 (16.2) | -3.2 (15.0)

23. Primary Outcome: Vital Signs- Sitting Diastolic Blood Pressure(DBP)
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 126 | 125
mmHg | -0.8 (11.2) | -1.3 (10.7)

24. Primary Outcome: Vital Signs- Pulse Rate
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 126 | 125
beats/minute | 3.2 (11.1) | 3.1 (11.5)

25. Primary Outcome: ECG Variables - Heart Rate
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 125 | 121
beats/minute | 3.6 (11.4) | 3.4 (10.9)

26. Primary Outcome: ECG Variables - QT Interval
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 125 | 121
ms | -4.5 (23.1) | -7.5 (21.2)

27. Primary Outcome: ECG Variables - QTcB Interval
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 125 | 121
ms | 3.6 (20.9) | 2.4 (22.6)

28. Primary Outcome: ECG Variables - QTcF Interval
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 125 | 121
ms | 0.7 (16.3) | -1.1 (17.4)

29. Primary Outcome: ECG Variables - RR Interval
Description: Change from baseline
Time Frame: Baseline and 52 week after
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 125 | 121
ms | -30.9 (121.4) | -43.8 (115.1)

30. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) symptoms_Night-time Awakening
Description: There are 5 alternatives (scored 0 to 4, 0= no awakening and 4 =did not sleep at all). The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period and daily during 52-week randomization treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 130 | 130
units on a scale | 0.0 (0.5) | -0.1 (0.4)

31. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) symptoms_Breathlessness
Description: There are 5 alternatives (scored 0 to 4, 0= unaware of any difficulty and 4 =almost constant, present even when resting). The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period and daily during 52-week randomization treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 130 | 130
units on a scale | -0.2 (0.7) | -0.1 (0.7)

32. Secondary Outcome: Chronic Obstructive Pulmonary Disease (COPD) symptoms_cough
Description: There are 5 alternatives (scored 0 to 4, 0= unaware of coughing, 4= never free of cough or need to cough). The change from Run-in period average to Treatment period average for each treatment group
Time Frame: Daily during run-in period and daily during 52-week randomization treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 130 | 130
units on a scale | -0.2 (0.7) | -0.2 (0.7)

33. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Measured With the Spirometer at the Clinic
Description: The ratio of the average value of available data for Weeks 0, 4, 8, 17, 26, 34, 43 and 52 to the baseline for each treatment group. Ratio is being reported as a percentage in this Measure.
Time Frame: Before randomization, 0, 4, 8, 17, 26, 34, 43 and 52 weeks after randomization
Measure: Geometric Mean (Full Range); unit: percentage of Baseline
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 129 | 129
percentage of Baseline | 104.25 [60.8 to 182.9] | 98.43 [35.8 to 168.2]

34. Secondary Outcome: Forced Vital Capacity (FVC) Measured With the Spirometer at the Clinic
Description: as for outcome 33
Time Frame: Before randomization, 0, 4, 8, 17, 26, 34, 43 and 52 weeks after randomization
Measure: Geometric Mean (Full Range); unit: percentage of Baseline
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 129 | 129
percentage of Baseline | 102.51 [77.8 to 141.5] | 100.04 [67.6 to 158.2]

35. Secondary Outcome: Time to First COPD Exacerbation
Description: A Chronic Obstructive Pulmonary Disease (COPD) exacerbation was defined as worsening in COPD symptoms requiring treatment with either a course of systemic steroid or hospitalisation. The percentage of participants who had experienced COPD exacerbation at the end of the study for each treatment group.
Time Frame: Daily during 52-week randomization treatment
Measure: Number; unit: Percentage of participants
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 130 | 130
Percentage of participants | 20.0 | 31.5

36. Secondary Outcome: Number of COPD Exacerbations Over the Study Treatment Period
Description: A Chronic Obstructive Pulmonary Disease (COPD) exacerbation was defined as worsening in COPD symptoms requiring treatment with either a course of systemic steroid or hospitalisation. Number of COPD exacerbation during 52-week randomization treatment
Time Frame: Daily during 52-week randomization treatment
Measure: Number; unit: event
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 130 | 130
event | 41 | 105

37. Secondary Outcome: Rescue Medication Use
Description: The change from run-in period and daily during 52-week randomization treatment
Time Frame: Daily during 52-week randomization treatment
Measure: Mean (Standard Deviation); unit: innhalation/day
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 130 | 130
innhalation/day | -0.2 (1.0) | 0.0 (1.4)

38. Secondary Outcome: Health Related Quality of Life (HRQL) Based on the St. George's Respiratory Questionnaire (SGRQ)
Description: The change from run-in period and daily during 52-week randomization treatment average for each treatment group. The SGRQ ranges from 0 (no impairment of quality of life) to 100 (highest impairment of quality of life).
Time Frame: Daily during run-in period and daily 52-week randomization treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 130 | 130
units on a scale | -2.03 (8.56) | -0.42 (7.47)

39. Secondary Outcome: Morning Peak Expiratory Flow (PEF) Measured at Home
Description: The change from Run-in period average to 52-week randomization Treatment period average for each treatment group
Time Frame: Daily during run-in period and daily 52-week randomization treatment
Measure: Mean (Standard Deviation); unit: Liter/minute(L/min)
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 126 | 123
Liter/minute(L/min) | 5.9 (31.8) | 5.7 (30.9)

40. Secondary Outcome: Evening Peak Expiratory Flow (PEF) Measured at Home
Description: The change from Run-in period average to 52-week randomization Treatment period average for each treatment group
Time Frame: Daily during run-in period and daily 52-week randomization treatment
Measure: Mean (Standard Deviation); unit: Liter/minute(L/min)
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 125 | 122
Liter/minute(L/min) | 2.7 (30.0) | 5.2 (29.3)

41. Secondary Outcome: Morning FEV1 Measured by the Subjects at Home
Description: The change from run-in period and daily during 52-week randomization treatment
Time Frame: Daily during run-in period and daily 52-week randomization treatment
Measure: Mean (Standard Deviation); unit: Liter(L)
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 126 | 123
Liter(L) | 0.017 (0.147) | 0.006 (0.171)

42. Secondary Outcome: Evening FEV1 Measured by the Subjects at Home
Description: The change from run-in period and daily during 52-week randomization treatment
Time Frame: Daily during run-in period and daily 52-week randomization treatment
Measure: Mean (Standard Deviation); unit: Liter(L)
Arm/Group | Arm 1 - Symbicort Turbuhaler | Arm 2 - COPD Standard Therapy
Number analyzed (Participants) | 125 | 122
Liter(L) | 0.006 (0.142) | 0.010 (0.156)

ADVERSE EVENTS:
Arm/Group | Symbicort Turbuhaler | COPD Standard Therapy
Serious Adverse Events (participants affected / at risk) | 25/130 | 34/130
Other Adverse Events (participants affected / at risk) | 75/130 | 72/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort Turbuhaler (N=130) | COPD Standard Therapy (N=130)
Arteriosclerosis Obliterans (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Prostatitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Benign Prostatic Hyperplasia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haematuria (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Computerised Tomogram Thorax Abnormal (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Inguinal Hernia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intervertebral Disc Protrusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Synovial Cyst (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Optic Ischaemic Neuropathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angle Closure Glaucoma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cataract (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Heat Illness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tendon Rupture (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Spinal Compression Fracture (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Syncope (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Loss Consciousness (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebral Infarction (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Prostate Cancer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Gastric Adenoma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal Cancer (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung Neoplasm Malignant (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary Tuberculosis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pneumonia Bacterial (Respiratory, thoracic and mediastinal disorders) | 0 | 5
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 20
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort Turbuhaler (N=130) | COPD Standard Therapy (N=130)
Insomnia (Psychiatric disorders) | 7 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Back Pain (Musculoskeletal and connective tissue disorders) | 6 | 10
Constipation (Gastrointestinal disorders) | 10 | 13
Pneumonia (Infections and infestations) | 9 | 3
Pharyngitis (Infections and infestations) | 9 | 3
Bronchitis (Infections and infestations) | 15 | 13
Nasopharyngitis (Infections and infestations) | 55 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other